CLINICAL TRIAL: NCT05070923
Title: Healthy Lifetime (HL): an Internet-based Behavioral Health Coaching Protocol for Older Adults
Brief Title: HealthyLifetime: Health Coaching for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Michigan Department of Health and Human Services (Other)
Responsible Party: Principal Investigator, Kathleen Potempa, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E20213681-001
Record Dates: First submitted 2021-09-23; First posted 2021-10-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Aging Well
Keywords: nurse coaching; motivational interviewing; aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HealthyLifetime Group (Experimental): HL is an 8-week, personalized health coaching program that includes a comprehensive assessment made through a survey and a "virtual' home visit (via video), a goal-directed strengthening action plan developed by the participant with the guidance of the nurse, a tailored daily planning guide to enhance action steps and goal attainment, and six weekly 30 minute nurse coaching sessions with participants the Healthie application technology via their personal home computer, Tablet or Smartphone device. If a participant does not use a personal device or the device cannot support the Healthie platform, the HL program will provide a Tablet to them for their use during the program. All video sessions ( ie, home visit, strengthening plan, and weekly coaching sessions will use a two-way video but only the audio portions of the sessions will be recorded. The HL program, tailored to each participant's need for strong and resilient function, encompasses the following key elements:
  Interventions: Behavioral: HealthyLifetime
- Usual Care Group (No Intervention): Participants randomized to the usual care group will be given information about when to expect reminders on the Healthie platform to complete future surveys at the end of week 8, and after three months that will be available on the Healthie Platform for them to fill out and save on the platform. They will also be reminded how to contact the study coordinator if they should have questions. Participants in this group will have the view to other functions on the platform turned off. They will only be able to view documents as the reminders appear for them to complete.

INTERVENTIONS:
Behavioral: HealthyLifetime — HL augments existing case management services by focusing on building the participant's personal capacity for independence in self - care skills, health behavior change, and health decision making. The HL program coordinates and interfaces with the enrollee's primary medical provider, case managers, and caregivers as necessary
  Arms: HealthyLifetime Group

SUMMARY:
To evaluate the benefits of the virtual 8-week program on selected health and functional outcomes, self-efficacy, and resiliency in a population over 50 years of age with one or more chronic conditions versus a randomized control group of like individuals.

DETAILED DESCRIPTION:
HL is an 8-week, personalized health coaching program that includes a comprehensive assessment made through a survey and a "virtual' home visit (via video), a goal-directed strengthening action plan developed by the participant with the guidance of the nurse, a tailored daily planning guide to enhance action steps and goal attainment, and six weekly 30 minute nurse coaching sessions with participants the Healthie application technology via their personal home computer, Tablet or Smartphone device. If a participant does not use a personal device or the device cannot support the Healthie platform, the HL program will provide a Tablet to them for their use during the program. All video sessions ( ie, home visit, strengthening plan, and weekly coaching sessions will use a two-way video but only the audio portions of the sessions will be recorded. The HL program, tailored to each participant's need for strong and resilient function, encompasses the following key elements:

Personal Health System Assessment (PHS Survey) - The foundational piece of HL is strengthening the participant's existing personal health system (PHS) - which we define as the network and interaction of an individual's strengths (such as beliefs, knowledge and skill for self-care and independence), social determinants of health, caregiver supports, and community resources, such as groceries, exercise, transportation, that the participant relies on to sustain health and function. The survey asks questions in the following domains: background information including income; social and spiritual network and support; personal health rating; use of healthcare services (emergency room visits, hospitalizations, primary care visits); lifestyle habits including use of tobacco, alcohol as well as diet, exercise, sleep and sexual behavior; health impact on activities, function, and symptoms; and self-efficacy in performing activities, in symptom management and in medication taking. The PHS Survey is completed by the participant through the web application and takes about 16 minutes to complete based on pilot data obtained in a sample of community living adults 50 years of age and older with one or more chronic conditions.

The PHS Survey results are reviewed by the UMSN Registered Nurse [either Advanced Practice Registered Nurse (APRN) or BSN- Prepared Registered Nurse (RN)] prior to the virtual home visit. During the virtual home visit, the nurse reviews the strengths of the PHS Survey, clarifies any information on the Medical History and conducts a home environment assessment completed by the participant under the guidance of the nurse. The nurse describes key results from the PHS Survey particularly focusing on their own words that describe their priority concerns and goals that they had expressed. The purpose of this is to maximize self-awareness and bring into focus the individual's own goals, strengths and areas for improvement forming the framework for beginning the PHS Plan process. The PHS Survey may reveal an individual's PHS network capacity (family, friends, community-organizations, church groups) to meet the person's need for additional in-home support for non-medical services such as housekeeping, bill paying, grocery shopping etc.

Personal Health System Strengthening Plan (PHS Plan) - The next step of the program includes creation of an individualized plan to strengthen capacity of the participant for self-care using the discussion of the PHS Survey and home assessments as a starting point for engaging the participant. The PHS Plan will be developed with the participant in a 45 - 60 minute video session the nurse. The PHS Plan assists the individual to set action steps to meet goals that reflect concerns about managing their medical regimen, medication taking, symptoms, daily living skills such as Activities of Daily Living (ADLs ) and Instrumental Activities of Daily Living (IADLs), and health behavior choices such as smoking, eating habits, activity etc. The nurse uses health coach motivational and nursing interviewing methods to support participant engagement, activation and self-efficacy in skills and decision-making. Goals and action steps progress throughout the 8-week program, with the guidance of the nurse, as the participant achieves success in reaching goals, making more independent choices, and gains self-care efficacy. By the conclusion of the HL program the participant is expected to have experienced the process of goal/action step/success so as to have sustaining capacity to continue the process without requiring the intensive support that HL provides.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older who have one or more chronic medical conditions (e.g., high blood pressure, diabetes, arthritis, obesity, etc.) which require management in some way (regular doctor checks, medication, etc.);
* Whose health is medically stable; that is, not currently undergoing either significant physical and/or mental health changes and not undergoing any type of non-routine treatments/medical testing or have any surgeries scheduled in the next six months;
* Has not had an ER visit related to his/her chronic conditions in the prior one month (an ER visit related to a one-time, resolved issue such as a bee sting or to have stitches for a household injury will not be cause for exclusion);
* Is able to read, speak and hear English; may use adaptive devices such as hearing aid and glasses;
* Is able to recall personal information such as age, DOB, address, phone number, and health history questions without difficulty;
* Reports having an established internet connection that is regularly used for video content [such as with Netflix, Amazon Prime, YouTube]; and
* Is able to use their internet connection in a private space.

Exclusion Criteria:

* Are acutely ill or have unstable health problems requiring medical work-up or follow-up clinic visits for monitoring more than every 3 months;
* Have had an ER visit related to his/her chronic condition in the prior one month; (an ER visit related to a one-time, resolved issue such as a bee sting or to have stitches for a household injury will not be cause for exclusion);
* Are terminally ill;
* Have severe memory problems;
* Have severe hearing and/or visual deficits that are not functionally adapted with devices such as a hearing aid or eye glasses;
* Do not have an existing internet connection at the bandwidth needed to support the video platform [cannot access video streaming content]; and/or
* Is able to use internet only in a public space (unable to ensure privacy).

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Change in Participant Self- rated health score | At 0, 8 and 12 weeks after study enrollment.
  Participants perception of their health on a scale of 1= Excellent to 5 = Poor
Change in Self-efficacy in ability to continue essential life activities score | At 0, 8 and 12 weeks after study enrollment.
  Confidence of the participant in doing certain activities on a scale of 1= Not at all confident to 10 = Totally Confident. For the purposes of answering these questions, confidence is defined as the belief in the participant's chances of being able to do and/or complete an activity (e.g., hobbies and recreation, social visits, chores, errands, etc.) or task (e.g., hobbies and recreation, social visits, chores, errands, etc.) successfully however the participant defines it.
Change in Independent self care agency score | At 0, 8 and 12 weeks after study enrollment.
  Confidence in doing certain activities, e.g., stick to behavior changes, meet goals, and improve health, on a scale of 1= Not at all confident to 10 = Totally Confident
Change in Health Habits score | At 0, 8 and 12 weeks after study enrollment.
  Activities that participants engage in that affect health in a negative or positive way, e.g., smoking (yes or no), alcohol (number of drinks per week), exercise (0 = none to 4= more than 3 hours/week), food choices (seldom or never to 2 or more times a day)
Change in Goal attainment score | At 0, 8 and 12 weeks after study enrollment.
  Health goals of participants (up to 3) and importance of goal (1= Not at all important now to 10 = highest importance now) and confidence in achieving goal (1= Not confident at all to 10 = Completely Confident)

SECONDARY OUTCOMES:
Change in Sustained higher values of primary measures at 3 months | 12 weeks after study enrollment
  Are effects of program noted at 8 weeks still present at 12 weeks.
Change in Self-reported medical visits | At 0, 8 and 12 weeks after study enrollment.
  Number of unplanned medical visits with doctor or primary medical provider in past 3 months (0 = no visits to 8 = 7 or more), emergency room visits (0 = none to 3 = 2 or more), overnight stay in hospital (0 = none to 3 = 2 or more).

OTHER OUTCOMES:
Change in Perception of health now and in 3 years score | At 0, 8 and 12 week after study enrollments.
  Participant thinks health now is and in three years will be 1 = Excellent to 5 = Poor.
Change in Level of Symptomatology score | At 0, 8 and 12 weeks after study enrollment.
  Frequency with which participants experience symptoms such as physical discomfort, pain, fatigue, etc. on a scale where 0 = Never to 5 = Always
Change in Confidence in ability to manage symptoms score | At 0, 8 and 12 weeks after study enrollment.
  How confident the participant is that they can keep health symptoms/problems from interfering with the things they want to do, e.g., fatigue, physical discomfort, emotional distress, etc. on a scale where 1 = Not at all Confident to 10 = Totally Confident
Change in Level of independence in activities score | At 0, 8 and 12 weeks after study enrollment.
  Ability to do daily living activities such as shopping, cooking, managing medications, etc. on a scale where 1 = Not at all Confident to 10 = Totally Confident
Change in Medication taking self care efficacy score | At 0, 8 and 12 weeks after study enrollment.
  Confidence of participants (on a scale where 0 = Not at all Confident to 2 = very Confident) in taking their medications correctly under different conditions, e.g., if take several medication each day, are away from home, if cause side effects, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Potempa, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan School of Nursing, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Potempa K, Calarco M, Flaherty-Robb M, Butterworth S, Marriott D, Potempa S, Laughlin C, Schmidt P, Struble L, Harden K, Ghosh B, Furspan P, Ellis A. A randomized trial of a theory-driven model of health coaching for older adults: short-term and sustained outcomes. BMC Prim Care. 2023 Oct 5;24(1):205. doi: 10.1186/s12875-023-02162-x. PMID 37798658